CLINICAL TRIAL: NCT01457313
Title: Comparison of Postoperative Pain in the First and Second Knee in Staged Bilateral Total Knee Arthroplasty: Clinical Evidence That Central Sensitization Increases Systemic Pain Sensitivity
Brief Title: Pain Compared Between the First and the Second Surgery in Staged BTKA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, Doctor, Seoul National University Bundang Hospital
Other Study IDs: TKA bilat pain
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BTKA: patients undergoing bilateral staged total knee arthroplasty

SUMMARY:
postoperative pain and analgesic consumption between the first and the second surgery would be compared in patients undergoing staged bilateral total knee arthroplasty (BTKA).

DETAILED DESCRIPTION:
postoperative pain and analgesic consumption is compared between the first and second total knee arthroplasty (TKA) operation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective bilateral staged total knee arthroplasty at a 1-week interval under spinal anesthesia,
* age <=85
* American Society of Anesthesiologists physical status of I to II

Exclusion Criteria: any contraindication to spinal anesthesia or femoral nerve block such as coagulopathy; conversion to general anesthesia; preexisting pain syndrome; abnormal liver function or renal test results; severe heart, liver, or renal disease; history of stroke or neurologic deficits; psychiatric disorder; chronic opioid use; drug dependency; allergy to study medications; inflammatory joint disease; previous surgery on or trauma of the knee; difference in preoperative VAS score of ≥ 20 (at rest and at maximum knee flexion) between each side of the knee; body mass index of ≥ 40 kg/m2; and inability to comprehend the VAS or to use patient-controlled analgesia (PCA.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing elective bilateral staged total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
VAS | from the end of the TKA surgery until postoperative 48 hour
  visual analogue scale

SECONDARY OUTCOMES:
analgesic consumption | from the end of the TKA surgery until postoperative 48 hour
  patient controlled analgesia (fentanyl)
rescue analgesic | from the end of the TKA surgery until postoperative 48 hour
  ketoprofen
antiemetics | from the end of the TKA surgery until postoperative 48 hour
  antiemetics total amount

CONTACTS AND LOCATIONS:
Overall Officials: Sanghwan Do, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hopital, Seongnam-si, Gyeonggi-do, South Korea